CLINICAL TRIAL: NCT07228650
Title: ADHD Remote Technology and ADHD Transition: Predicting and Preventing Negative Outcomes
Acronym: ART-transition
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other); South West London and St George's Mental Health NHS Trust (Other); Northamptonshire Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 334427
Record Dates: First submitted 2025-01-23; First posted 2025-11-14 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-01

CONDITIONS: Attention Deficit Hyerpactivity Disorder
Keywords: ADHD; attention-deficit/hyperactivity disorder; remote measurement technology; mHealth; Adolescence; medication adherence; Longitudinal
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescents with ADHD
- Informant: Parent or guardian of the individuals with ADHD

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) is a common neurodevelopmental condition affecting 5.9% of young people. Late adolescence can be a particularly challenging period for young people with ADHD, with major life transitions, new demands and increased expectations. This vulnerable phase also coincides with the transition from child and adolescent mental health care to adult ADHD services, where new UK data show that most young people with ADHD do not successfully transfer to adult services. Therefore, many young people with ADHD do not receive appropriate interventions at a time when they may need them most. Opportunities for intervention are currently not fully realised due to both the young people's disengagement from clinical services and our limited understanding of real-world targets for more holistic interventions. The current study seeks to address these needs using remote (not in-person) measurement technology (RMT). The MRC-funded project, ART-transition, will use the ADHD Remote Technology ('ART') assessment and monitoring assessments with young people with a diagnosis of ADHD aged 16-17 and the RADAR-base mobile-health platform to which it is linked. ART consists of active (e.g. questionnaires) and passive (e.g. sleep) smartphone app monitoring. In the study, the investigators will address three questions on the transition to adulthood for individuals with ADHD: what changes take place, what predicts them, and how can the investigators prevent negative outcomes and support healthy lifestyles? The investigators will remotely monitor 250 young people with ADHD over two years. The investigators will then co-design, with young people with ADHD, a prototype for a new ADHD-transition smartphone app. Our approach focuses on giving young people with ADHD greater autonomy in how they manage their ADHD, in collaboration with their clinician, and places the emphasis on modifiable environmental factors and the prevention of negative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DSM-5 ADHD
* Aged 16-17
* Able to give informed consent for participation
* Willing and able to complete self-reported assessments via smartphone
* Willing to use either their own compatible Android phone or a study Android - phone as their only smartphone during the data collection period
* Willing to wear the wearable device during the data collection period

Exclusion criteria

* Psychosis, currently experiencing a major depressive episode, mania, drug dependence in the last six months, or a major neurological disorder.
* Recent contact with psychiatric acute care (admission, crisis team or liaison team (A&E) in the last six months
* Any other major medical disease which might impact upon the patient's ability to participate in normal daily activities (e.g., due to hospitalisations)
* Pregnancy
* IQ < 70

Informant Inclusion Criteria:

* A parent or guardian, as chosen by the participant with ADHD
* Aged 18 or over
* Willing and able to complete web-based questionnaires regarding the participant with ADHD

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Community and secondary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
ADHD symptoms and functional impairment | Baseline and every 4 weeks up to month 24
  Barkley Adult ADHD Rating scale on symptoms and functional impairment (BAARS-IV)- Self Report. 29 items. For 18 items, individuals report the frequency with which they have experienced ADHD symptoms over the past two weeks on a four-point Likert Scale (0 = 'Never' or 'Rarely', 1 = 'Sometimes', 2 = 'Often', 3 = 'Very Often'). One item asks individuals to indicate the ages at which they first experienced symptoms. For the final 10 items, individuals report the extent to which their symptoms have interfered with their ability to function in various domains (e.g., home life or at work) on a four-point Likert Scale (0 = 'Never or Rarely', 1 = 'Sometimes', 2 = 'Often', 3 = 'Very Often').
ADHD symptoms | Baseline and every day up to month 24
  Non-validated daily ADHD symptom question. 1 item. Individuals report the extent to which ADHD symptoms affected their daily activities on a Likert Scale (1 = Not at all, 2 = Slightly, 3 = Somewhat, 4 = Quite a lot, 5 = A lot).
Anxiety (General Anxiety Disorder-7, GAD-7) | Baseline and every 4 weeks up to month 24
  7-items. 4-point Likert scale indicating the frequency of experiencing items in the past two weeks (0 = 'Not at all', 1 = 'Several days', 2 = 'More than half the days', 3 = 'Nearly every day'). Higher scores indicate higher severity of anxiety symptoms.
Depression (Patient Health Questionnaire -8, PHQ-8, adapted) | Baseline and every 4 weeks up to month 24
  8-items. 4-point Likert scale indicating the frequency of experiencing items in the past two weeks (0 = 'Not at all', 1 = 'Several days', 2 = 'More than half the days, 3 = 'Nearly every day'). Higher scores indicate higher severity of depression symptoms.
Aggression (Reactive-Proactive Aggression Questionnaire for Adults. RPQ-A, adapted) | Baseline and every 4 weeks up to month 24
  23 items, 3-point Likert scale rated from 0 to 2 (0 = 'Never', 1 = 'Sometimes', 2 = 'Often'), indicating the frequency of experiencing items in the past two weeks. Higher scores indicate increased aggression.
Irritability - (Affective Reactivity Index self-report, ARI-s, adapted) | Baseline and every 4 weeks up to month 24
  7-item, 3-point Likert Scale rated from 0 to 3 (0 = 'Not True', 1 = 'Somewhat True', 2 = 'Certainly True') indicating frequency of experiencing symptoms in the past two weeks.
Nicotine Dependence - The Fagerstrom Test for Nicotine Dependence | Baseline and every 4 weeks up to month 24
  6-items. Four items are yes/no questions rated from 0 to 1, and two are multiple-choice questions rated from 0 to 3 on a 4-point Likert scale. A higher score is associated with more nicotine dependence.
Alcohol Use (Alcohol Use Disorders Identification Test questionnaire, AUDIT) | Baseline and every 4 weeks up to month 24
  10 items, with a 4-point Likert scale rated from 0 to 3. A higher score is associated with more harmful or hazardous drinking.
Eating Disorders (Short Form of the Eating Disorder Examination Questionnaire, EDE-QS) | Baseline and every 6 months up to month 24
  12 items. 10 items are questions about behaviours in the past seven days, rated on a scale from 0 to 3 for frequency (0 = 0 days, 1 = 1-2 days, 2 = 3-5 days, 3 = 6-7 days). 2 items are about self-perception over the past seven days, rated on a scale from 0 to 3 for extent (0 = Not at all, 1 = Slightly, 2 = Moderately, 3 = Markedly). A higher score is associated with more eating disorder behaviours.
Self-esteem (Rosenberg Self-Esteem Scale, RSES) | Baseline and every 6 months up to month 24
  10 items. 4-point Likert scale format ('Strongly Agree', 'Agree', 'Disagree, 'Strongly Disagree'). Responses are assigned 1-4 points. Higher scores indicate higher self-esteem.
Social support and engagement with work/studies | Baseline and every 4 weeks up to month 24]
  Non-validated questionnaire
Healthy lifestyle behaviours and digital signals associated with changes in clinical symptoms | Continuously across a 24-month time period
  Passive monitoring using the RADAR-BASE smartphone "Passive App" measuring digital signals of behaviour.
Healthy lifestyle behaviours and digital signals associated with changes in clinical symptoms | Continuously across a 24-month time period
  Passive monitoring using a Fitbit wearable device measuring sleep. Device sensors, including an accelerometer and a photoplethysmographic pulse oximeter, will be combined to calculate sleep duration.
Healthy lifestyle behaviours and digital signals associated with changes in clinical symptoms | Continuously across a 24-month time period
  Passive monitoring using a Fitbit wearable device measuring physical activity. Device sensors, including a gyroscope and an accelerometer, will be combined to calculate step count.
Markers associated with clinical symptoms - cognitive measures | Baseline and every 6 months up to month 24
  Continuous Performance Test/Go No-Go Task (Combined Task)
Markers associated with clinical symptoms - cognitive measures | Baseline and every 6 months up to month 24
  Fast Task

CONTACTS AND LOCATIONS:
Overall Officials: Jonna Kuntsi, PhD, Principal Investigator — Social, Genetic and Developmental Psychiatry Centre, Institute of Psychiatry, Psychology and Neuroscience, King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not relevant

REFERENCES:
- See also: RADAR-base mobile-health platform developed by Dobson et al. — http://www.radar-base.org
- See also: ADHD Remote Technology ('ART') assessment and monitoring assessments developed by Kuntsi, Dobson, et al. — https://www.kcl.ac.uk/research/adhd-remote-technology-art